CLINICAL TRIAL: NCT00618358
Title: A Prospective, Randomized, Multi-Center, Two Arm Study to Evaluate the Safety and Effectiveness of the Vascular Sealant System Compared With Gelfoam/Thrombin for Control of Anastomosis Suture Line Bleeding in Patients Undergoing Vascular Reconstructive Surgery With PTFE Grafts
Brief Title: Vascular Sealant Study
Acronym: VSS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor - Confluent Surgical terminated study re: surgical techniques Letter dated 4/31/2008
Sponsor: Georgetown University (Other)
Collaborators: Medtronic - MITG (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007-072
Record Dates: First submitted 2008-02-08; First posted 2008-02-20 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2010-01

CONDITIONS: Arteriovenous Access Grafts or Extra-anatomic and Infra-inguinal Grafts
MeSH Terms: interventions — Gelatin Sponge, Absorbable; Thrombin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vascular Sealant) (Experimental)
  Interventions: Device: Vascular Sealant System
- Gelfoam/Thrombin (Active Comparator)
  Interventions: Other: Gelfoam/Thrombin

INTERVENTIONS:
Device: Vascular Sealant System — The Vascular Sealant System is intended for use in vascular reconstructions to achieve adjunctive hemostasis by mechanically sealing areas of leakage.
  Arms: Vascular Sealant)
Other: Gelfoam/Thrombin
  Arms: Gelfoam/Thrombin

SUMMARY:
Study Objective:To evaluate the safety and effectiveness of the Vascular Sealant compared with Gelfoam/Thrombin when used to seal bleeding anastomotic suture lines in patients undergoing vascular reconstructive surgery requiring placement of a PTFE graft (including extra-anatomic, infrainguinal bypass and arteriovenous (AV) access procedures).

Study Design: The study is a multi-center, prospective, randomized controlled clinical trial that will compare two methods for treating anastomotic leakage (bleeding). All subjects (n =151) will be randomized at a 3:1 ratio to receive either the investigational treatment (Vascular Sealant) or the control treatment (Gelfoam/Thrombin). Up to two (2) treatment sites may be evaluated for each subject. Subjects will be stratified by type of graft procedure: AV access graft or extra-anatomic and infra-inguinal graft. A minimum of 60 patients, and a maximum of 91 patients, will be enrolled in each stratum. Treatment randomization will be blocked by center and type of graft procedure (e.g., bypass or AV grafts). All subjects will undergo preoperative screening to determine eligibility and will be evaluated intraoperatively, at discharge or within 7 days of surgery, and 30 days post-procedure to monitor for hematologic disturbances, hemorrhagic events, wound complications and other potential acute post-operative adverse events.

Up to ten (10) investigational sites will participate in the study. Enrollment is expected to take approximately 8 months for an anticipated duration of the clinical investigation of approximately 9 to 10 months.

The primary objective of this trial is to demonstrate non-inferiority of the Vascular Sealant to Gelfoam/Thrombin when used to seal anastomotic suture lines in patients undergoing placement of PTFE vascular grafts (including extra-anatomic, infrainguinal bypass and arteriovenous access procedures).

ELIGIBILITY:
Preoperative Inclusion Criteria:

Subjects must meet all of the following criteria to be eligible for participation in the study:

* > 18 years of age
* Scheduled for elective vascular surgery that entails placement of a PTFE vascular graft including extra-anatomic, infrainguinal bypass and primary and secondary arteriovenous access procedures
* Subject is willing and able to comply with all aspects of the treatment and evaluation schedule
* Informed of the nature of the study, and has provided written informed consent, approved by the appropriate Institutional Review Board (IRB) of the respective clinical site

Preoperative Exclusion Criteria: Subjects who meet any of the following criteria are not eligible for participation in the study:

* Subject has a known local or systemic infection
* Subjects with known coagulapathies including hemophilia, factor deficiencies, platelet count < 80,000 u/mL, heparin induced thrombocytopenia or uncorrected INR > 1.5
* Subject is participating in a clinical trial that requires treatment with another investigational device or drug
* Subject is lactating or pregnant, or does not agree to use contraception for the duration of the study
* Subject has a known hypersensitivity to any components of bovine thrombin preparations and/or material of bovine origin
* The investigator determines that the subject should not be included in the study for reason(s) not already specified

Intraoperative Inclusion Criteria: Subjects must meet the following intraoperative inclusion criteria to be eligible for randomization:

• Suture line leaks (bleeding) confirmed prior to randomization.

Intraoperative Exclusion Criteria: Subjects who meet any of the following intraoperative exclusion criteria are considered screening failures and are not eligible to be randomized:

* Incidental finding of any of the preoperative exclusion criteria
* Subject has obvious contamination or a concurrent systemic infection
* Investigator determines that participation in the study may jeopardize the safety or welfare of the subject

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2007-03

CONTACTS AND LOCATIONS:
Overall Officials: David Deaton, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Ma GW, Kucey A, Tyagi SC, Papia G, Kucey DS, Varcoe RL, Forbes T, Neville R, Dueck AD, Kayssi A. The role of sealants for achieving anastomotic hemostasis in vascular surgery. Cochrane Database Syst Rev. 2024 May 2;5(5):CD013421. doi: 10.1002/14651858.CD013421.pub2. PMID 38695613